CLINICAL TRIAL: NCT05984524
Title: Gamma-Music Based Intervention for Mild Alzheimer's Disease
Acronym: NUGammaMBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NortheasternMINDLabGammaMBI
Record Dates: First submitted 2023-06-16; First posted 2023-08-09 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Masking Description: Sham placebo control intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamma (Experimental): 8-week music-based intervention with gamma lights
  Interventions: Behavioral: Gamma-Music Based Intervention
- Control (Placebo Comparator): 8-week music-based intervention with control lights
  Interventions: Behavioral: Gamma-Music Based Intervention

INTERVENTIONS:
Behavioral: Gamma-Music Based Intervention — Gamma or Control lights with Music-Based Intervention for 8 week period

SUMMARY:
The study will test and refine a novel brain-stimulation tool using gamma-frequency lights coupled with self-selected music for a gamma-music-based intervention for participants with mild Alzheimer's Disease. Results will yield a gamma-stimulation protocol that reliably influences brain activity (Aim 1), is adaptive, motivating and rewarding to use (Aim 2), and will generate predictions as to who might benefit the most from gamma-MBI (Aim 3). By bridging the gap between neurostimulation and behavioral intervention by combining music therapy with gamma- band neurostimulation, the present project aims to find a sustainable intervention that delays the progression of AD.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is characterized by cognitive deficits such as memory loss, as well as deficits in the motivation that drives daily activities. These cognitive and motivational deficits are linked to widespread neuronal and synaptic atrophy, coupled with aggregated extracellular Aβ-plaque and tau deposits, and atypical neural activity across multiple frequencies. Recent work in mouse models of AD have shown that inducing gamma oscillations with a non-invasive gamma-frequency (40 Hz) light-flickering and auditory tone-stimulation regimes reduced Aβ plaques and improved spatial and recognition memory. In humans, restoring gamma-frequency activity while preserving its phase-amplitude coupling with theta-band activity are shown to recover human memory performance in older adults, and in patients with mild AD, thus offering a promising route towards a novel therapy that can prevent brain atrophy while improving cognition. Despite their recent successes, it is a major challenge to translate gamma-frequency neurostimulation from a laboratory study to a behavioral intervention. The goal is to promote healthy neurocognitive aging using lifestyle interventions; in particular, interventions that sustainably elevate mood and reward motivated behavior while encouraging social bonding may be most promising in slowing the progression of AD. Music listening engages multiple brain networks involved in sensory processing, movement, language, attention, learning and memory, emotion and reward, and social connectedness. Music-Based Interventions (MBIs) have the potential to manage symptoms, slow disease progression, and improve quality of life. This study will test a novel protocol for music-based brain stimulation, gamma-MBI: gamma-light stimulation that automatically adapts to music-based intervention. Harnessing the fact that music listening is an intrinsically rewarding activity, the study uses music as a carrier for gamma sensory stimulation. As music contains theta-band acoustic energy, music listening is a form of theta- band noninvasive brain stimulation. A novel brain-stimulation tool will be tested using gamma-frequency lights coupled with self-selected music for a gamma-music-based intervention for participants with mild Alzheimer's Disease. Results will yield a gamma-stimulation protocol that reliably influences brain activity (Aim 1), is adaptive, motivating and rewarding to use (Aim 2), and will generate predictions as to who might benefit the most from gamma-MBI (Aim 3). By bridging the gap between neurostimulation and behavioral intervention by combining music therapy with gamma-band neurostimulation, the present project aims to find a sustainable intervention that delays the progression of AD.

ELIGIBILITY:
Mild AD participants will be ages 55-90, amnestic (single or multiple domain) who perform below an education- adjusted cut-off score on the Logical Memory II subscale delayed paragraph recall of the Wechsler Memory Scale-Revised (WMS-R LM-IIa) (Wechsler 1987) (≥16 years: ≤8; 8-15 years: ≤4; 0-7 years: ≤2), have a CDR global score of 0.5 (with a memory box score of 0.5 or 1), have an MMSE score of 20-24, and have preserved instrumental activities of daily living (ADL) as determined by the Alzheimer's Disease Cooperative Study ADL Prevention Instrument (ADCS ADL-PI). All participants will be medically stable. Participants will not have significant cerebrovascular disease determined by history of stroke, and will have a Modified Hachinski Ischemic score (Rosen et al. 1980) of ≤ 4. Participants will not have significant psychiatric disorders including a Geriatric Depression Scale (long form) (Yesavage et al. 1982) of ≤10, and will not have a history of substance or alcohol abuse. All participants must be on stable doses of any medications with psychotropic effects (including cholinesterase inhibitors, memantine, and antidepressants) for at least 3 months prior to randomization. Participants will be screened to be amyloid positive via plasma test. They must also have no contraindications to MRI scanning, and will have a study partner who is able to provide collateral information about the participant. A pure tone audiogram will be administered to ensure that participants have no more than mild levels of hearing loss (<40dB). If a subject fails audiometric screening, they will be excluded from the study and provided with a list of audiologists. An Institutional Review Board (IRB) approved telephone screen will be used for demographic information, study inclusion/exclusion criteria and MRI contraindications. Participants will complete an MRI screening questionnaire before each MRI session.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
EEG activity | 1 hour
  Gamma-band EEG activity

SECONDARY OUTCOMES:
ADAS-Cog 14 | 8 weeks
  cognitive component of iADRS

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided